CLINICAL TRIAL: NCT03397797
Title: Effect of Intraoperative Neuromuscular Blockade on Postoperative Sore Throat and Hoarseness in Patients Undergoing Spinal Surgery
Brief Title: Effect of Intraoperative Neuromuscular Blockade on Postoperative Sore Throat and Hoarseness
Status: Completed | Type: Observational
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, associate professor, SMG-SNU Boramae Medical Center
Other Study IDs: 20170605/10-2017-6/063
Record Dates: First submitted 2017-11-09; First posted 2018-01-12 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Sore Throat
Keywords: muscle relaxant
MeSH Terms: conditions — Pharyngitis; Muscle Hypotonia | interventions — Rocuronium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group with muscle relaxant: Rocuronium is used during the operation to maintain moderate relaxation.
  Interventions: Drug: Rocuronium
- Group without muscle relaxant: Rocuronium is not used during the operation for the eletrophysiological monitoring.

INTERVENTIONS:
Drug: Rocuronium — In the group to need the eletrophysiological monitoring during the operation, we don't inject muscle relaxant except anestheitic induction.
  Groups: Group with muscle relaxant

SUMMARY:
Investigators assess and compare postoperative sore throat and hoarseness in the group using the muscle relaxant and not using it during the operation.

DETAILED DESCRIPTION:
The muscle relaxant is usually used during the operation to maintain moderate relaxation but, it can't be used in the surgery to need eletrophysiological monitoring during the operation. In this sturdy, the investigators assess the postoperative sore throat and hoarseness and compare the effect of muscle relaxant in the group using the muscle relaxant and not using it in terms of the incidence and severity of postoperative sore throat and hoarseness.

ELIGIBILITY:
Inclusion criteria

* patients scheduled to undergo elective lumbar spinal surgery Exclusion criteria
* known or predicted difficult airway
* neuromuscular diseases
* hepatic or renal dysfunction
* diseases or anatomical abnormalities in the neck, larynx, or pharynx
* requirement for postoperative mechanical ventilation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for elective lumbar spinal surgery
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Overall cumulative incidence of postoperative sore throat | Within 24 hr evaluation period after operation
  The incidence sore throat is assessed by the presence of sore throat
Overall cumulative incidence of postoperative hoarseness | Within 24 hr evaluation period after operation
  The incidence sore throat is assessed by the degree of hoarseness

SECONDARY OUTCOMES:
Incidence of postoperative sore throat | At 1,6, and 24 hr after operation
  The incidence of sore throat is assessed by the presence of sore throat.
Severity of postoperative sore throat | At 1,6, and 24 hr after operation
  A 0-100 mm NRS is used to evaluate the severity of sore throat (0, no pain; 100, worst pain imaginable).
Incidence and severity of postoperative hoarseness | At 1,6, and 24 hr after operation
  Hoarseness is defined as a voice quality different from the preoperative voice and graded as follows: none (no hoarseness), mild (recognized by the patient), moderate (obvious to the investigator), and severe (aphonia).
Post operative analgesic consumption | within 24 hrs after operation
  the amount of patient-controlled analgesia and other analgesic medication consumed

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Yong Hwang, M.D.,Ph. D., Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Jee-Eun Chang, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No